CLINICAL TRIAL: NCT04266899
Title: The Effect of Neuro-orthosis on Gait Performer in Chronic Post Stroke Subjects
Brief Title: The Effect of Neuro-orthosis on Gait Performer in Post Stroke Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Aline de Souza Pagnussat, Principal Investigator, Federal University of Health Science of Porto Alegre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FDS_Stroke
Record Dates: First submitted 2020-01-28; First posted 2020-02-12 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Stroke
Keywords: Cerebrovascular Stroke; Cerebral Stroke; Cerebrovascular Accident; Neurorehabilitation; Gait Rehabilitation
MeSH Terms: conditions — Stroke | interventions — Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FDS+Treadmill gait training (Experimental): Chronic stroke patients submitted to Foot Drop Stimulation (FDS) + Treadmill gait training during two weeks.
  Interventions: Device: Foot Drop Stimulator - Neuro Orthosis; Device: Treadmill

INTERVENTIONS:
Device: Foot Drop Stimulator - Neuro Orthosis — The WalkAide system is a self-contained functional electrical stimulation device with a built-in tilt sensor and attaches with a cuff to the leg below the knee. The device stimulates the peroneal nerve provides active dorsiflexion of muscle during the swing phase of gait.
Device: Treadmill — Gait training on a treadmill

SUMMARY:
The aim of this study is to verify the effectiveness of foot drop stimulation (FDS) on gait rehabilitation of post-stroke subjects with mild, moderate and severe compromise.

DETAILED DESCRIPTION:
The stroke subjects are going to perform the walking training with Foot drop stimulator on the treadmill. All the evaluations will be performed with a foot drop stimulator turned off and on. One month later, that finished the intensive treatment; the participants were also evaluated only without the stimulation of FDS.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with ischemic or hemorrhagic stroke diagnosis.
* Mild, moderate or severe hemiparesis (chronic stroke - at least 6 months)
* Minimal cognitive ability to understand commands
* Able to walk 10 meters unassisted or with minimal assistance

Exclusion Criteria:

* Secondary musculoskeletal disorder involving the lower limb
* Contraindication for electrical stimulation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-09-20 (Actual); Primary Completion 2019-09-20 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
Assessment of gait speed | Change from Pre to Post treatment (2 weeks) and Post 3 (1 month follow-up)
  Evaluated by means of the 3-D motion analysis system (capture system BTS SMART DX 400)

SECONDARY OUTCOMES:
Assessment of angular kinematics of hip, knee and ankle | Change from Pre to Post treatment (2 weeks) and Post 3 (1 month follow-up)
  Evaluated by means of the 3-D motion analysis system (capture system BTS SMART DX 400)
Changes in center of pressure displacement | Change from Pre to Post treatment (2 weeks) and Post 3 (1 month follow-up)
  Assessed by force platform (BTS P-6000)
Postural Control | Change from Pre to Post treatment (2 weeks) and Post 3 (1 month follow-up)
  Evaluated by Center of Pressure (COP) displacement assessed on force platform (BTS P-6000)
Functional Mobility | Change from Pre to Post treatment (2 weeks) and Post 3 (1 month follow-up)
  Evaluated by means of the Timed Up & Go Test (TUG)
Muscular tone assessed by the Modified Ashworth Scale | Change from Pre to Post treatment (2 weeks) and Post 3 (1 month follow-up)
  Assessed by the Modified Ashworth Scale. This scale consists of 5 ordinal values ranging from 0 (no tonus increase) to 4 (stiffness).
Assessment of Sensorimotor Recovery After Stroke by Fugl-Meyer scale | Change from Pre to Post treatment (2 weeks) and Post 3 (1 month follow-up)
  Fugl-Meyer scale of lower limb impairment. The evaluation includes measurement of voluntary movement, velocity, coordination and reflex activity, through an ordinal scale applied to each item: 0- cannot be performed, 1- partially performed, and 2-performed completely. Participants were also classified according their LL motor impairment in severe (0 to19), moderate (20 to 28) or mild (> 29 points).
Assessment of Gait speed in external environment | Change from Pre to Post treatment (2 weeks) and Post 3 (1 month follow-up)
  Evaluated by means inertial sensor (G-Sensor®, BTS Bioengineering, Italy) during 10 meters walking test.
Assessment of duration of stance and swing phase of gait | Change from Pre to Post treatment (2 weeks) and Post 3 (1 month follow-up)
  Evaluated by means inertial sensor (G-Sensor®, BTS Bioengineering, Italy), during 10 meters walking test.
Assessment of Stride length and Step length of gait | Change from Pre to Post treatment (2 weeks) and Post 3 (1 month follow-up)
  Evaluated by means inertial sensor (G-Sensor®, BTS Bioengineering, Italy), during 10 meters walking test.
Assessment of cadence by means number of steps by the minute. | Change from Pre to Post treatment (2 weeks) and Post 3 (1 month follow-up)
  Evaluated by means inertial sensor (G-Sensor®, BTS Bioengineering, Italy), during 10 meters walking test.
Assessment of Harmonic Ration of Gait | Change from Pre to Post treatment (2 weeks) and Post 3 (1 month follow-up)
  Evaluated by means single miniaturized inertial sensor (G-Sensor®, BTS Bioengineering, Italy). The device collects the values of linear accelerations along three orthogonal axes (antero-posterior (AP) corresponding to the walking direction, medio-lateral (ML), and supero-inferior (V)). The Harmonic Ration is the ratio between the sum of the amplitudes of even harmonics and the sum of the amplitudes of odd harmonics calculated via the discrete Fourier transform along the antero-posterior (AP) and cranio-caudal (CC) directions; the opposite ratio is calculated along the latero-lateral axis (LL).

CONTACTS AND LOCATIONS:
Overall Officials: Aline S Pagnussat, PhD, Principal Investigator — Federal University of Health Sciences of Porto Alegre
Locations (1):
- Federal University of Health Sciences of Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil